CLINICAL TRIAL: NCT06229119
Title: Vault Evaluation After Implantation of an Implantable Collamer Lens
Brief Title: Vault Evaluation After ICL Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 23-003
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-01

CONDITIONS: Nearsightedness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: All subjects were implanted with the EVO ICL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ICL (Other): ICL implantation
  Interventions: Device: Implantable Collamer Lens

INTERVENTIONS:
Device: Implantable Collamer Lens — The EVO ICL lens is intended to be placed entirely within the posterior chamber directly behind the iris and in front of the anterior capsule of the human crystalline lens. When correctly positioned, the EVO ICL lens functions as a refractive element to optically reduce moderate to high myopia with or without astigmatism.

SUMMARY:
The purpose of this study is to evaluate the lens vault after implantation of an implantable collamer lens (ICL). The ICL is designed to be implanted in front of the eye, without removing the natural lens. Because of this, it is also known as a phakic IOL. The ICL has already been approved by the U.S. Food and Drug Administration (FDA) to treat mid to high degrees of refractive errors such nearsightedness (also called myopia) with or without astigmatism. Once the artificial lens is implanted, a space between the ICL and the crystalline lens is created, which is called vault.

DETAILED DESCRIPTION:
The ICL will be implanted in both eyes of study subjects. Diagnostic instrumentation will be used to measure the vault between the ICL and the crystalline lens.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Males and Females.
* Age: 21 to 45 years of age
* Willing and able to provide written informed consent for participation in the study
* Willing and able to comply with scheduled visits and other study procedures.
* Scheduled to undergo ICL implantation in both eyes within 1 to 30 days between surgeries.
* Subjects who require an ICL power in the range of -3.00 to -15.00 D.

Exclusion Criteria:

* Patients who do not qualify for an ICL according to the Direction For Use (DFU)
* Unstable or worsening myopia
* Use of any systemic or topical drug known to interfere with visual performance.
* Irregular astigmatism.
* History of retinal detachment.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
* Pigment dispersion
* Previous intraocular surgery.
* Previous refractive surgery.
* Previous keratoplasty
* Pupil abnormalities
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Solomon, MD, Principal Investigator — Carolina Eyecare Physicians
Locations (1):
- Helga Sandoval, Mt. Pleasant, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was expected to be 33 per the protocol, but enrollment proved difficult. 21 subjects were screened, with one screen failure. Twenty subjects started and completed the study.
Units Other Than Participants: Eyes
Groups:
- ICL Implantation Group: ICL implantation
  Implantable Collamer Lens: The EVO ICL lens is intended to be placed entirely within the posterior chamber directly behind the iris and in front of the anterior capsule of the human crystalline lens. When correctly positioned, the EVO ICL lens functions as a refractive element to optically reduce moderate to high myopia with or without astigmatism.
Period: Overall Study
Arm/Group | ICL Implantation Group
Started | 20; 40 Eyes
Completed | 20; 40 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | ICL Implantation Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference Between Predicted and Actual Central Vault at 1-month After ICL Implantation
Description: Difference between the predicted vault at the preoperative visit and the actual vault measured at the 1-month visit
Time Frame: 1-month
Population: Patients with ICL placed horizontally were included in the analysis.
Measure: Mean (Standard Deviation); unit: Milimeters
Units Other Than Participants: eyes
Arm/Group | ICL Implantation Group
Number analyzed (Participants) | 15
Number analyzed (eyes) | 30
Milimeters | 0.170 (0.137)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | ICL Implantation Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT06229119/Prot_SAP_000.pdf